CLINICAL TRIAL: NCT01433848
Title: Prospective Analysis Of Cardiac Function In Cirrhotic Patients By Echocardiography And Its Correlation With Adverse Events
Brief Title: Prospective Analysis Of Cardiac Function In Cirrhotic Patients By Echocardiography And Its Correlation With Events
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Angelo Antunes Salgado, Clinical practitioner, Rio de Janeiro State University
Other Study IDs: arquivo1
Record Dates: First submitted 2011-08-09; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Child A liver cirrhosis
- Child B liver cirrhosis
- Child C liver cirrhosis

SUMMARY:
The cardiac abnormalities in patients with cirrhosis are already reported from the 50's, in studies of patients with alcoholic cirrhosis. Further studies have shown that these cardiac changes were caused not only by the myotoxic effects of alcohol, but also are present in many patients regardless of etiology of cirrhosis.

These changes are characterized by abnormalities of systolic contraction in patients undergoing physical or pharmacological stress, changes in diastolic function and electrophysiological changes in a clinical condition known as cirrhotic cardiomyopathy. Increased QT interval and the pre-ejection time changes are common in cirrhotic patients.

To date no studies have evaluated the clinical relevance of changes in the heart of cirrhotic patients, or their relationship with the prognosis of affected patients. Til now, researches are based on strict echocardiographic parameters, not including several modern methods of assessment of cardiac systole and diastole. New techniques, such as two-dimensional strain, can bring new diagnostic and prognostic information, and it is not reported in the literature. Therefore, the aim of this study is to determine the morphological and functional cardiac changes in patients with cirrhosis and their prognostic role by evaluating new echocardiographic parameters of systolic and diastolic readings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis of any etiology, diagnosed by clinical criteria and ultrasound and / or liver biopsy, which excluded patients with causes that also may affect cardiac function (hemochromatosis, Wilson disease, amyloidosis).
* Age between 18 and 80 years.
* Signing of written informed consent.

Exclusion Criteria:

* History or presence of systemic arterial hypertension (treated or not)
* History or presence of ischemic heart disease and peripheral vascular disease.
* Presence of greater than mild valvular disease.
* Patients who have a different rhythm in the baseline electrocardiogram, other than sinus (atrial fibrillation, atrial flutter, junctional rhythm).
* Presence of severe anemia (Hb <7 g / dL).
* Presence of shock, hepatic encephalopathy, bacterial infection or bleeding at inclusion or during the previous week.
* History or presence of severe or decompensated lung disease.
* Presence of percutaneous intrahepatic porto-systemic shunt (TIPS).
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Will be selected patients with cirrhosis (diagnosed by clinical criteria and ultrasound and / or liver biopsy) at different evolutionary stages os disease in the hepatology's service at the University Hospital Pedro Ernesto.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Adverse events as defined as composite of death due to liver failure, gastrointestinal bleeding, spontaneous bacterial peritonitis or need to conduct liver transplant in patients with liver cirrhosis. | 12 months follow-up
  Identify the occurrence of adverse events as defined as:
  1. death due to liver failure, characterized by development of severe liver injury with impaired synthetic function and encephalopathy in a person who previously had well-compensated liver disease.
  2. either upper or lower gastrointestinal bleeding, characterized by hematemesis (vomiting of blood or coffee-ground like material) and/or melena (black, tarry stools).
  3. spontaneous bacterial peritonitis, characterized by as an ascitic fluid infection without an evident intraabdominal surgically-treatable source.
  4. liver transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo A Salgado, Master, Principal Investigator — Rio de Janeiro State University; Carlos Terra, PHD, Study Chair — Rio de Janeiro State University; Márcia B Castier, PHD, Study Chair — Rio de Janeiro State University; Paulo R Benchimol-Barbosa, DSC, Study Chair — Rio de Janeiro State University; Camila SS Reis, MD, Principal Investigator — Universidade de Estado do Rio de Janeiro
Locations (1):
- Universidade do Estado do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Salgado AA, Barbosa PRB, Ferreira AG, Reis CASS, Terra C. Prognostic Value of a New Marker of Ventricular Repolarization in Cirrhotic Patients. Arq Bras Cardiol. 2016 Dec;107(6):523-531. doi: 10.5935/abc.20160181. PMID 28558079